CLINICAL TRIAL: NCT00486265
Title: A Phase I/II, Open-Label, Multi-Center, Two-Part Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of AZD4877 Administered on Days 1, 2 and 3 in Adult Patients With Recurrent or Refractory Acute Myelogenous Leukemia (AML) Excluding Promyelocytic Leukemia
Brief Title: Phase I/II, Open-label, Multi-center, Two Part Dose-escalation, Safety, Pharmacokinetics (PK) and Efficacy Study of AZD4877 in Patients With Acute Myelogenous Leukemia (AML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: AML assess. of response in Part B patients find treatment failure in all 8 evaluable for marrow response following a maximum of 2 induction courses of therapy
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2782C00007
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Results first posted 2010-08-17 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-07

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Phase I; Phase II; acute myelogenous leukemia; AML; cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — N-(3-aminopropyl)-N-(1-(5-benzyl-3-methyl-4-oxo-(1,2)thiazolo(5,4-d)pyrimidin-6-yl)-2-methylpropyl)-4-methylbenzamide

INTERVENTIONS:
Drug: AZD4877 — intravenous infusion administered on days 1, 2 and 3

SUMMARY:
The primary purpose of this study is to find out what the maximum tolerated dose is for an experimental drug called AZD4877 based on the side effects experienced by patients that receive AZD4877 on a daily times 3 schedule in acute myelogenous leukemia (AML).

For enrollment information see the Central Contact information below

ELIGIBILITY:
Inclusion Criteria:

* Part A: Relapsed or refractory leukemia for which no standard therapies are anticipated to result in a durable remission
* Part B: AML who have had no more than two prior relapses or failed to achieve remission after at least one induction treatment.
* Patients with prior allogeneic transplants who remain clinically stable for ≥2 weeks or more off immunosuppressive therapy

Exclusion Criteria:

* Promyelocytic acute myelogenous leukemia
* Prior allogeneic transplant requiring immunosuppressive therapy or treating physician does not consider patient to be a candidate for allogeneic transplantation.
* Liver injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-07; Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Curt, MD, Study Director — AstraZeneca
Locations (4):
- United States (3):
  - Research Site, Chicago, Illinois
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
- Research Site, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kantarjian HM, Padmanabhan S, Stock W, Tallman MS, Curt GA, Li J, Osmukhina A, Wu K, Huszar D, Borthukar G, Faderl S, Garcia-Manero G, Kadia T, Sankhala K, Odenike O, Altman JK, Minden M. Phase I/II multicenter study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD4877 in patients with refractory acute myeloid leukemia. Invest New Drugs. 2012 Jun;30(3):1107-15. doi: 10.1007/s10637-011-9660-2. Epub 2011 Apr 15. PMID 21494838

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 4 study sites in the United States and 1 study site in Canada between July 2007 and February 2009 [Part A] and between March 2009 and July 2009 [Part B].
Pre-assignment Details: Following enrolment there was screening period of up to 28 days, after which if all inclusion/exclusion criteria were met, patients were dosed with AZD4877
Groups:
- AZD4877: AZD4877 [ Time Frame: administered on days 1,2 and 3]
Period: Overall Study
Arm/Group | AZD4877
Started | 9 (Partipants dosed on day 1.)
Completed | 0 (Treatment is not for a fixed period and continues until a discontinuation criterion is met)
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 8

BASELINE CHARACTERISTICS:
Arm/Group | AZD4877
Number analyzed (Participants) | 9
Age, Customized [Number; unit: Participants]
  < 18 Years | 0
  >=18 - < 65 Years | 6
  >=65 - < 75 Yrs | 1
  >=75 Yrs | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 8
  Black or African American | 1

OUTCOME MEASURES:

1. Primary Outcome: To Identify a Maximum Tolerated Dose (MTD) of AZD4877 by Assessment of the Incidence of Dose-limiting Toxicities (DLTs)
Description: To identify a maximum tolerated dose (MTD) of AZD4877 by assessment of the incidence of dose-limiting toxicities (DLTs)
Time Frame: Dose-limiting toxicities (DLTs) are evaluated during the first induction treatment course administered during the initial 15-day treatment period.
Reporting Status: Not Posted
Measure: Number; unit: Participants

2. Primary Outcome: To Assess the Effect of AZD4877 on the Rate of Complete Remission (CR)
Description: Marrow response is assessed by modified Cheson criteria for Acute Myelogenous Leukemia (AML). Possible outcomes for marrow response are CR (Complete Remission), CRi (Complete Remission with incomplete blood count recovery), PR (Partial Remission), and treatment failure.
Time Frame: Response is evaluated after a maximum of 2 courses of induction therapy.
Population: 8 of 9 patients in Part B were evaluable for response following a maximum of 2 courses of induction therapy.
Measure: Number; unit: Participants
Arm/Group | AZD4877
Number analyzed (Participants) | 8
Participants | 0

3. Primary Outcome: To Determine the PK Profile of AZD4877 [ Time Frame: Daily x 3 Schedule ]
Description: Maximum plasma concentration, Cmax
Time Frame: PK samples are collected on Days 1, 2, 3, 24 and 48 hours following the end of Day 3 AZD4877 infusion and Day 8.
Reporting Status: Not Posted
Measure: Geometric Mean (Standard Deviation); unit: ng/mL

4. Secondary Outcome: To Assess the Effect of AZD4877 on Rate and Duration of CR, CRi, PR and Overall Response (CR,CRi, or PR)
Description: as for outcome 2
Time Frame: Response is evaluated after a maximum of 2 courses of induction therapy.
Reporting Status: Not Posted
Measure: Number; unit: Participants

5. Secondary Outcome: To Evaluate the Safety and Tolerability of AZD4877 on a Daily x 3 Schedule by Assessment of Adverse Events, Non-hematologic Labs and Vital Signs
Time Frame: Patients were followed for safety from the date of first dose of AZD4877 up to 30-days after the last administration of AZD4877, where possible.
Reporting Status: Not Posted
Measure: Number; unit: Participants

ADVERSE EVENTS:
Arm/Group | AZD4877
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD4877 (N=9)
Mucosal Inflammation (General disorders) | 3
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD4877 (N=9)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Hypophosphatasia (Congenital, familial and genetic disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Dry Eye (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Mucosal Inflammation (General disorders) | 6
Fatigue (General disorders) | 3
Oedema Peripheral (General disorders) | 2
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Oedema (General disorders) | 1
Hepatic Cyst (Hepatobiliary disorders) | 1
Hepatic Lesion (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Ear Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Limb Injury (Injury, poisoning and procedural complications) | 1
Transfusion Reaction (Injury, poisoning and procedural complications) | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 1
Blood Phosphorus Increased (Investigations) | 1
Blood Pressure Orthostatic Decreased (Investigations) | 1
Transaminases Increased (Investigations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3
Decreased Appetite (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1
Haemangioma Of Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 3
Neuropathy Peripheral (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Mood Altered (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal Cyst (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
On 16 June 2009, the study was terminated for a lack of efficacy. None of the 8 patients had experienced CR or CRi. The secondary efficacy outcome measures were not evaluated due to early termination and small number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to provide a copy of the publication to AZ for review at least 60 days in advance of submission for publication. Investigators in multicenter (MC) studies agree to postpone MC publications until the earlier of the date of the first AZ authorized MC publication or a period up to 18 months from study completion at all sites. AZ has the right to request delays: up to 60 days for confidential information, and an additional 90 days to protect intellectual property.